CLINICAL TRIAL: NCT00768690
Title: A Study in Healthy Adult Subjects to Evaluate the Safety, Tolerability, and Pharmacokinetics of Multiple Doses of ABT-333
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Daniel Cohen, MD/Study Medical Director, Abbott
Allocation: Randomized | Model: Single Group | Masking: Triple
Other Study IDs: M10-687
Record Dates: First submitted 2008-10-07; First posted 2008-10-08 (Estimated); Last update posted 2010-10-13 (Estimated); Status verified 2010-09

CONDITIONS: HCV Infection
MeSH Terms: conditions — Hepatitis C | interventions — dasabuvir; Ketoconazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (5):
- 1 (Other): Healthy volunteers, receiving daily doses of 200 mg ABT-333 or placebo, BID for 10 days; and on Study Day 11 receiving a single dose of 200 mg ABT-333 or placebo + 400 mg ketoconazole
  Interventions: Drug: ABT-333; Drug: ketoconazole; Drug: placebo
- 2 (Other): Healthy volunteers, receiving 400 mg ABT-333 or placebo, BID
  Interventions: Drug: ABT-333; Drug: placebo
- 3 (Other): Healthy volunteers, receiving 600mg ABT-333 or placebo, BID
  Interventions: Drug: ABT-333; Drug: placebo
- 4 (Other): Healthy volunteers, receiving 1000mg ABT-333 or placebo, BID
  Interventions: Drug: ABT-333; Drug: placebo
- 5 (Other): Healthy volunteers, receiving 1600mg ABT-333 or placebo, BID*
  *After review of the data from previous groups, and in accordance with the protocol, this arm was not dosed.
  Interventions: Drug: ABT-333; Drug: placebo

INTERVENTIONS:
Drug: ABT-333 — Capsule, or powder drug substance from the capsule powder mixed in an alternate vehicle. For additional information refer to arm description.
Drug: ketoconazole — Tablet, see arms for intervention description
  Arms: 1
Drug: placebo — Capsule or powder drug substance from the capsule powder mixed in an alternative vehicle. For additional information refer to arm description.

SUMMARY:
The purpose of this study is to determine multiple dose safety, tolerability and pharmacokinetics of ABT-333 under nonfasting conditions in healthy adult subjects, and to determine the effect of single dose administration of ketoconazole on steady state ABT-333 pharmacokinetics

DETAILED DESCRIPTION:
Phase 1, Blinded, Randomized, Placebo-controlled Study in Healthy Adult Subjects to Evaluate the Safety, Tolerability, and Pharmacokinetic Profiles of Multiple Doses of ABT-333

ELIGIBILITY:
Inclusion Criteria:

* Main Selection Criteria for Healthy Volunteers:

  * Subject has provided written consent.
  * Subject is in general good health.
* If female, subject is postmenopausal for at least 2 years or surgically sterile.
* If female, subject is not pregnant and is not breast-feeding.
* Male or female between 18 and 55 years old, inclusive.
* If male, subject must be surgically sterile or practicing at least 1 method of birth control.
* Body Mass Index (BMI) is 18 to 29, inclusive.

Exclusion Criteria:

* See above for main selection criteria

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2008-10; Primary Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Analysis of pharmacokinetic results. | Approximately 1 week.
Analysis of safety measures including but not limited to tabulation of adverse events, physical exam, clinical lab results (include chemistry, hematology and urine) and vital signs. | Approximately 1 week.

SECONDARY OUTCOMES:
Analysis of single dose administration of ketoconazole on steady state ABT-333 pharmacokinetics. | Approximately 1 week.

CONTACTS AND LOCATIONS:
Locations (1):
- Site Reference ID/Investigator# 12701, Waukegan, Illinois, United States